CLINICAL TRIAL: NCT00070473
Title: A Phase I Study of Pemetrexed (LY231514, Alimta) in Children and Adolescents With Recurrent Solid Tumors
Brief Title: Pemetrexed Disodium in Treating Young Patients With Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ADVL0311; NCI-04-C-0261 (Other: NCI Trial Identifier); CDR0000334572 (Other: Clinical Trials.gov); COG-ADVL0311 (Other: Children's Oncology Group)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium, use different ways to stop tumor cells from dividing so they stop growing or die. Pemetrexed disodium may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase I trial is studying the side effects and best dose of pemetrexed disodium in treating young patients with recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of pemetrexed disodium in children and adolescents with refractory solid tumors.
* Determine the dose-limiting toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

Secondary

* Determine, preliminarily, the antitumor activity of this drug in these patients.
* Correlate the presence of the C677T polymorphism of the methylenetetrahydrolate reductase gene, the presence of a polymorphism in the enhancer region of the thymidylate synthase (TS) gene promoter (2R and 3R tandem repeats), the presence of a polymorphism within one of those repeats, and the presence of a functional polymorphism in the 3'-untranslated region with toxicity in patients treated with this drug.
* Correlate homocysteine and methylmalonic acid levels at study entry with toxicity in patients treated with this drug.
* Correlate various gene expression profiles with response in patients treated with this drug.

OUTLINE: This is a dose-escalation study.

Patients receive pemetrexed disodium IV over 10 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of pemetrexed disodium until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 3-36 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor for which there is no known curative therapy or therapy that is known to prolong survival with acceptable quality of life

  * Histologic requirement waived for intrinsic brain stem tumors
* No pleural effusion or ascites
* Neurological deficits from CNS tumors must have been relatively stable for at least 1 week prior to study entry

PATIENT CHARACTERISTICS:

Age

* 1 to 21

Performance status

* Karnofsky 50-100% (over 10 years of age)
* Lansky 50-100% (10 years of age and under)

Life expectancy

* At least 8 weeks

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 8.0 g/dL (transfusion allowed)

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 2.5 times ULN
* Albumin at least 2 g/dL

Renal

* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min OR
* Creatinine based on age as follows:

  * No greater than 0.8 mg/dL (age 5 and under)
  * No greater than 1.0 mg/dL (age 6 to 10)
  * No greater than 1.2 mg/dL (age 11 to 15)
  * No greater than 1.5 mg/dL (age 16 and over)

Pulmonary

* No evidence of dyspnea at rest
* No exercise intolerance

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No evidence of Approved-not yet active graft-versus-host disease
* No uncontrolled infection
* Seizure disorder allowed provided it is well-controlled with anticonvulsants
* CNS toxicity no greater than grade 1

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy
* At least 7 days since prior antineoplastic biologic therapy
* At least 6 months since prior allogeneic stem cell transplantation
* More than 1 week since prior growth factors
* No concurrent biologic therapy
* No concurrent immunotherapy
* No concurrent prophylactic growth factor support during course 1

Chemotherapy

* No prior pemetrexed disodium
* More than 3 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No other concurrent chemotherapy

Endocrine therapy

* Concurrent dexamethasone for CNS tumors allowed provided dose has been stable or decreasing for at least 1 week prior to study entry

Radiotherapy

* Recovered from all prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy
* At least 6 months since prior craniospinal radiotherapy
* At least 6 months since prior radiotherapy to 50% or more of the pelvis
* At least 6 weeks since prior substantial bone marrow radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No trimethoprim or sulfa within 2 days before and after study drug administration
* No concurrent nonsteroidal anti-inflammatory agents (e.g., ibuprofen and aspirin)
* No other concurrent anticancer or investigational agents

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2003-10; Primary Completion 2006-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | Length of study

SECONDARY OUTCOMES:
Dose Limiting Toxicity | Length of study
  Any patient who experiences DLT at any time during protocol therapy will be considered evaluable for toxicity. Patients not experiencing DLT must complete a full cycle of therapy to be considered potentially evaluable for toxicity. Patients who are not evaluable for toxicity will be replaced.
Maximum Tolerated Dose | Length of study
  The MTD will be that dose at which fewer than one-third of patients experience DLT

CONTACTS AND LOCATIONS:
Overall Officials: H. Stacy Nicholson, MD, MPH, Study Chair — OHSU Knight Cancer Institute; Linda C. Stork, MD, Study Chair — Doernbecher Children's Hospital at Oregon Health and Science University
Locations (20):
- United States (18):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - NCI - Pediatric Oncology Branch, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Fairview University Medical Center - University Campus, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec

REFERENCES:
- [Result] Malempati S, Nicholson HS, Reid JM, Blaney SM, Ingle AM, Krailo M, Stork LC, Melemed AS, McGovern R, Safgren S, Ames MM, Adamson PC; Children's Oncology Group. Phase I trial and pharmacokinetic study of pemetrexed in children with refractory solid tumors: the Children's Oncology Group. J Clin Oncol. 2007 Apr 20;25(12):1505-11. doi: 10.1200/JCO.2006.09.1694. PMID 17442992